CLINICAL TRIAL: NCT07073326
Title: Effects of Normobaric Hypoxia Aerobic Training in People With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Brief Title: Effects of Normobaric Hypoxic Training in Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Acronym: HYPOMASLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Alex Buoite Stella, PhD, Assistant Professor, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DSM_FisioMedSport_Hypoxic25
Record Dates: First submitted 2025-06-01; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Normobaric Hypoxia
Keywords: Hypoxia; Altitude; Exercise; Liver; Metabolism; Fat
MeSH Terms: conditions — Hypoxia; Motor Activity; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYPOTRAIN (Experimental): This arm will perform the normobaric hypoxic aerobic training (HYPOTRAIN)
  Interventions: Other: HYPOTRAIN
- NORMOTRAIN (Sham Comparator): This arm will perform the normobaric normoxia aerobic training (NORMOTRAIN)
  Interventions: Other: NORMOTRAIN

INTERVENTIONS:
Other: HYPOTRAIN — 8 weeks of 2/3 times per week, 1-h aerobic training (walking on a treadmill at 60-65% HRmax) while wearing a mask and air is delivered between 15 and 16 FiO2%
  Arms: HYPOTRAIN
Other: NORMOTRAIN — 8 weeks of 2/3 times per week, 1-h aerobic training (walking on a treadmill at 60-65% HRmax) while wearing a mask and air is delivered between at normal (around 21) FiO2%
  Arms: NORMOTRAIN

SUMMARY:
Altitude training has been suggested to be of potential support to improve some chronic clinical conditions, especially metabolic conditions. Normobaric hypoxia represents a promising system to simulate altitude training, and its efficacy and safety have been suggested in different conditions, including diabetes, obesity and hypertension. Metabolic dysfunction-associated steatotic liver disease (MASLD) can characterized by metabolic alterations (including altered body composition, lipid and glycemic profile, etc.), and might benefit from aerobic training performed in simulated altitude training (i.e., normobaric hypoxia). Mild altitude training will be proposed (equal to about 2'500 m, 15% FiO2) and compared to a sham normobaric normoxia condition, during an 8-week 3 or 2 times per week 1-h aerobic training (walking) at 60-65% of maximum heart rate (HRmax). Cardiorespiratory fitness, body composition, and metabolic profile will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MASLD from at the least 3 years
* BMI > 26 kg/m2
* Being sedentary

Exclusion Criteria:

* Cardiovascular, respiratory, renal complications
* Hypertension
* COPD
* Previous history of acute mountain sickness or altitude-associated symptoms
* Females only: pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Body mass (kg) | At the beginning of the study and after 8 weeks of training
  Evaluation of changes in body mass measured on a scale
Fat mass (%) | At the beginning of the study and after 8 weeks of training
  Evaluation of changes in fat mass, as percentage of body mass, assessed with bioimpedence (BIA)

SECONDARY OUTCOMES:
Maximum oxygen uptake (mL/kg*min) | At the beginning of the study and potentially after 8 weeks of training
  Maximum oxygen uptake (VO2 max) assessed during a cardiopulmonary exercise test (CPET)
Liver markers | At the beginning of the study and after 8 weeks of training
  Markers of liver health including ultrasound evaluation
Ventilatory threshold (mL/kg*min) | At the beginning of the study and potentially after 8 weeks of training
  Metabolic intensity at which the ventilatory threshold occurs, as measured during the cardiopulmonary exercise test (CPET)
Triglyceride (mg/dL) | At the beginning of the study and after 8 weeks of training
  Blood triglyceride concentration
Total cholesterol (mg/dL) | At the beginning of the study and after 8 weeks of training
  Blood total cholesterol concentration
High-density lipoprotein (mg/dL) | At the beginning of the study and after 8 weeks of training
  Blood high-density lipoprotein concentration
Low-density lipoprotein (mg/dL) | At the beginning of the study and after 8 weeks of training
  Blood low-density lipoprotein concentration
C-reactive protein (mg/dL) | At the beginning of the study and after 8 weeks of training
  Blood c-reactive protein concentration
Glycemia (mg/dL) | At the beginning of the study and after 8 weeks of training
  Blood glucose concentration
Insulinemia (mg/dL) | At the beginning of the study and after 8 weeks of training
  Blood insulin concentration

REFERENCES:
- [Background] Luo Y, Chen Q, Zou J, Fan J, Li Y, Luo Z. Chronic Intermittent Hypoxia Exposure Alternative to Exercise Alleviates High-Fat-Diet-Induced Obesity and Fatty Liver. Int J Mol Sci. 2022 May 6;23(9):5209. doi: 10.3390/ijms23095209. PMID 35563600
- [Background] DE Groote E, Britto FA, Bullock L, Francois M, DE Buck C, Nielens H, Deldicque L. Hypoxic Training Improves Normoxic Glucose Tolerance in Adolescents with Obesity. Med Sci Sports Exerc. 2018 Nov;50(11):2200-2208. doi: 10.1249/MSS.0000000000001694. PMID 29923910